CLINICAL TRIAL: NCT01358383
Title: A Phase I, Open-label, Single-center Study to Assess the Pharmacokinetics of a Single Oral Dose of VIMOVO (250 mg Naproxen/20 mg Esomeprazole)in Healthy Adult Subjects
Brief Title: Assessment of Pharmacokinetics of a Single Oral Dose of VIMOVO in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D1120C00040
Record Dates: First submitted 2011-05-16; First posted 2011-05-23 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: Juvenile Idiopathic Arthritis; Pharmacokinetics; VIMOVO; fasting state; Amount of VIMOVO in the blood; taken on empty stomach
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Naproxen; Esomeprazole

INTERVENTIONS:
Drug: naproxen — 250mg, oral dose
Drug: esomeprazole — 20mg, oral dose

SUMMARY:
This is an assessment of Pharmacokinetics of a single oral dose of VIMOVO in healthy adult volunteers.

DETAILED DESCRIPTION:
A Phase I, Open-label, Single-center Study to Assess the Pharmacokinetics of a Single Oral Dose of VIMOVO (250 mg Naproxen/20 mg Esomeprazole)in Healthy Adult Subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects aged 18 to 55 years
* Capable of understanding and complying with the Clinical Study Protocol
* Body mass index (BMI) of 19 to 30 kg/m2 and weight of 50 to 100 kg

Exclusion Criteria:

* Previous enrollment in the present study
* Receipt of another investigational product within 4 weeks before this study or plans to participate in another study at the same time as this study
* Female subjects with a positive urine pregnancy test

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2011-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Observed maximum concentration (Cmax) | Pharmacokinetic samples will be collected at pre-dose, 10, 20, 30, and 45 minutes post-dose, and 1, 1.5, 2,2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours post-dose. The 72 hour post-dose sample will be collected at Visit 3 (Follow-up).
time of maximum concentration (tmax) | Pharmacokinetic samples will be collected at pre-dose, 10, 20, 30, and 45 minutes post-dose, and 1, 1.5, 2,2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours post-dose. The 72 hour post-dose sample will be collected at Visit 3 (Follow-up).
area under the concentration-time curve from zero to time of last quantifiable concentration (AUC(0-t)) | Pharmacokinetic samples will be collected at pre-dose, 10, 20, 30, and 45 minutes post-dose, and 1, 1.5, 2,2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours post-dose. The 72 hour post-dose sample will be collected at Visit 3 (Follow-up).
area under the concentration-time curve from zero to infinity (AUC) | Pharmacokinetic samples will be collected at pre-dose, 10, 20, 30, and 45 minutes post-dose, and 1, 1.5, 2,2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours post-dose. The 72 hour post-dose sample will be collected at Visit 3 (Follow-up).
apparent terminal rate constant (λz), apparent terminal half-life (t1/2) | Pharmacokinetic samples will be collected at pre-dose, 10, 20, 30, and 45 minutes post-dose, and 1, 1.5, 2,2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours post-dose. The 72 hour post-dose sample will be collected at Visit 3 (Follow-up).
apparent systemic clearance after extravascular dosing (CL/F) | Pharmacokinetic samples will be collected at pre-dose, 10, 20, 30, and 45 minutes post-dose, and 1, 1.5, 2,2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours post-dose. The 72 hour post-dose sample will be collected at Visit 3 (Follow-up).
apparent volume of distribution following extravascular dosing (Vz/F) for naproxen and esomeprazole | Pharmacokinetic samples will be collected at pre-dose, 10, 20, 30, and 45 minutes post-dose, and 1, 1.5, 2,2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours post-dose. The 72 hour post-dose sample will be collected at Visit 3 (Follow-up).

SECONDARY OUTCOMES:
Incidence and severity of Adverse events during the study as a measure of safety and tolerability | Collected from administration of VIMOVO (Visit 2 [Residential period] Day 1) until the end of the study, including follow-up
Abnormalties in Clinical laboratory tests (hematology, clinical chemistry, and urinalysis) as a measure of safety and tolerability | Labs will be taken from screening to follow up visit
Abnormalities in Vital signs as a measure of safety and tolerability | From screening to follow up visit

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sostek, Study Director — AstraZeneca; Bo Fransson, Study Chair — AstraZeneca; Kelly Craven, Principal Investigator — Quintiles Phase I Services, Overland Park, Kansas
Locations (1):
- Research Site, Overland Park, Kansas, United States